CLINICAL TRIAL: NCT00998621
Title: Development and Validation of a Questionnaire Measuring Treatment Adherence in Patients With Hepatitis C
Brief Title: ADHEPTA Study: Adherence Questionnaire in Hepatitis C
Acronym: ADHEPTA
Status: Completed | Type: Observational
Sponsor: Fundacion IMIM (Other)
Responsible Party: Sponsor
Other Study IDs: ADH-HEPC-2009-01
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Hepatitis C, Chronic; HIV Infection
Keywords: Hepatitis C, Chronic; HIV Infection; Medication Adherence; Questionnaire Design; Treatment experienced
MeSH Terms: conditions — Hepatitis C, Chronic; HIV Infections; Medication Adherence

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hepatitis C infection
  Interventions: Other: Adherence questionnaire
- Hepatitis C + HIV infections
  Interventions: Other: Adherence questionnaire

INTERVENTIONS:
Other: Adherence questionnaire — Adherence questionnaire

SUMMARY:
Main objective: To study and validate a questionnaire measuring treatment adherence in patients with Hepatitis C virus (HCV) infection.

Design of the study: Multicentric, prospective, epidemiological study in the field of usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patient infected by HCV according to diagnosis criteria used en usual clinical practice.
* Patient no treated previously and beginning a treatment for HCV.
* Patient that signed the informed consent to participate in the study.
* Group A: patient with HCV monoinfection.
* Group B: patient with HCV and HCV co-infection (according to diagnosis criteria used en usual clinical practice).

Exclusion Criteria:

* Patient that received previous treatment for HCV.
* Patient that is going to participate in a clinical trial Turing the HCV treatment period.
* Patient with cognitive impairment or patient unable to understand and answer the auto-administered questionnaire.
* Patient unable to read or write Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCV and with HCV + HIV
Sampling Method: Non-Probability Sample
Enrollment: 1120 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Main objective of the study is the development and validation of a Questionnaire measuring treatment adherence in patients with HCV infection. | 2 years

SECONDARY OUTCOMES:
Adherence will be measured according to 80/80/80 rule. | 2 years
Establish a relationship between adherence, virological response (VR) and Sustained virological response (SVR). | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain